CLINICAL TRIAL: NCT03052140
Title: Post-approval Study to Assess Lamelleye vs Comparator for the Treatment of Dry Eye Disease in Adults
Brief Title: Lamelleye vs Comparator for the Treatment of Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: Lamellar Biomedical Ltd (Industry); University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 001170
Record Dates: First submitted 2016-10-11; First posted 2017-02-14 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A, followed by Treatment B (Other): Treatment group that will receive Treatment A for 14 days, followed by Treatment B for 14 days. There will be a minimum 7 day washout between Treatments. Lamelleye Dry Eye Drops and Optive Plus will be administered to all subjects in this arm. Treatments will be self-administered at least 3 times a day.
  Interventions: Device: Lamelleye Dry Eye Drops; Device: Optive Plus
- Treatment B, followed by Treatment A (Other): Treatment group that will receive Treatment B for 14 days, followed by Treatment A for 14 days. There will be a minimum 7 day washout between Treatments. Lamelleye Dry Eye Drops and Optive Plus will be administered to all subjects in this arm. Treatments will be self-administered at least 3 times a day.
  Interventions: Device: Lamelleye Dry Eye Drops; Device: Optive Plus

INTERVENTIONS:
Device: Lamelleye Dry Eye Drops — Liposomal multi-dose preservative-free sterile suspension which contains soy lecithin phospholipids, sphingomyelin and cholesterol, suspended in saline.
  Other Names: CXB/1-14
Device: Optive Plus — Multi-dose sterile solution which contains sodium carboxymethylcellulose, glycerine, Castor Oil, Polysorbate 80, levocarnitine, and erythritol, preserved with PURITE® which breaks down into natural tear components in the eye

SUMMARY:
Single-blind, randomised, single centre, 2-way crossover study to collect post-market clinical follow-up data on the CE-marked Lamelleye dry eye drops medical device.

DETAILED DESCRIPTION:
The study is a 2-way crossover design comprising 2 treatments: the CE-marked Lamelleye dry eye drops, and a CE-marked comparator product. All Participants will be allocated to a treatment group in a random order.

This study design allows observations to be made between the treatments at both an intra- and inter-patient level regarding relationships between the patients' disease specific quality of life, symptoms and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written informed consent.
2. Male or female Participants ≥ 18 and ≤ 79 years of age.
3. Participant has dry eye disease as diagnosed from positive responses to Non-invasive tear break-up time (NITBUT) (≤10 seconds); Schirmer test (≤10mm in 5 minutes); and patient symptoms (>2 symptoms using the McMonnies Dry Eye Questionnaire)
4. Participant must understand and be able, willing and likely to fully comply with study procedures and restrictions.

Exclusion Criteria:

1. Active ocular infection
2. Ocular surgery within 6 months of study start date
3. Current contact lens wear
4. Any ophthalmologic drops within 1 week prior to enrolment that in the opinion of the CI or PI may interfere with the study outcomes.
5. Started or changed the dose of chronic systemic medication known to affect tear production including, but not limited to antihistamines, anticholinergics, antidepressants, diuretics, corticosteroids or immunomodulators within 30 days of initial visit.
6. Systemic disease known to affect tear production or loss including, but not limited to thyroid eye disease, that has been diagnosed or has not been stable within 30 days of Visit 1.
7. Known hypersensitivity to any of the agents used in testing such as allergies to egg or soya based products.
8. Females who are or wish to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Non-invasive tear break-up time (outcome used to power study) | 14 days (analysed for each Treatment period)
  Measure of time taken from blink to breakup of tear film

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | 14 days (analysed for each Treatment period)
  12-item questionnaire designed to assess the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning
Symptom Assessment in Dry Eye (SANDE) | 14 days (analysed for each Treatment period)
  Two questions which each use a horizontal visual analogue technique to quantify patient symptomatology of dryness and/or irritation
Evaporimetry | 14 days (analysed for each Treatment period)
  Measure of the rate of evaporation of the tear film from the surface of the eye.
Interferometry | 14 days (analysed for each Treatment period)
  Tear film lipid layer interferometry is a test to study the structure and quality of the lipid layer in the tear film.
Osmolarity | 14 days (analysed for each Treatment period)
  Tear osmolarity is a test to determine the solute concentration of the tear film.
Corneal and Conjunctival Staining | 14 days (analysed for each Treatment period)
  Corneal and conjunctival damage due to dry eye can be measured by staining the surface of the eye with fluorescein and examining under a lamp with a cobalt blue filter

CONTACTS AND LOCATIONS:
Overall Officials: Ian Pearce, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available